CLINICAL TRIAL: NCT04019834
Title: Preoperative Regional Nerve Block to Decrease Acute and Chronic Post-Operative Pain and Narcotic Use Following Mastectomy
Brief Title: Preoperative Regional Nerve Block for Acute and Chronic Post-Operative Pain Following Mastectomy
Acronym: RELIEF
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rachael Lancaster, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-300003680
Record Dates: First submitted 2019-04-03; First posted 2019-07-15 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Mastectomy; Anesthesia, Local; Narcotic Use
MeSH Terms: conditions — Breast Neoplasms | interventions — Steroids; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients and all study and hospital personnel will be blinded to randomization assignments except the regional anesthesia team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- regional nerve block with local anesthesia (Experimental): Treatment Arm (n=55) will receive titrated sedation with a combination of fentanyl and versed prior to the start of the block. An ultrasound will be used to identify the fascial planes and perform regional nerve blocks. A block needle will be passed into the fascial plane an injectate will be deposited . The injectate in the active arm will contain a local anesthestic and dexamethasone.
  Interventions: Drug: regional nerve block with local anesthesia of bupivacaine with steroid
- regional nerve block with normal saline (Placebo Comparator): Placebo Comparator Arm (n=55). Patients will undergo the same procedure with the exception of injection of 10cc of normal saline into the subcutaneous tissue.
  Interventions: Other: Placebo regional nerveblock with normal saline

INTERVENTIONS:
Drug: regional nerve block with local anesthesia of bupivacaine with steroid — Patient will receive titrated sedation with a combination of fentanyl and versed prior to the start of the block. An ultrasound will be used to identify the fascial planes for either pectoral, serratus, or erector spinae nerve blocks. A block needle will be passed into the fascial plane and injectate will be deposited. The injectate in the active arm will contain a combination of bupivacaine, epinephrine and dexamethasone.
  Other Names: Bupivicaine
  Arms: regional nerve block with local anesthesia
Other: Placebo regional nerveblock with normal saline — Patients who are randomized to placebo will undergo the same procedure with the exception of injection of 10cc of normal saline into the subcutaneous tissue .
  Other Names: Placebo
  Arms: regional nerve block with normal saline

SUMMARY:
The purpose of this study is to see if pre-operative regional nerve blocks compared to a placebo nerve block can decrease chronic post mastectomy pain, immediate postoperative pain and postoperative narcotic consumption.

DETAILED DESCRIPTION:
Surgical intervention of breast cancer is vital to breast cancer treatment or prevention and patient outcomes. However, surgical therapy can lead to chronic pain that may affect quality of life for breast cancer survivors including the potential for long-term disability. Chronic pain after breast cancer surgery is common, occurring in about 25-50% of patients. This chronic pain commonly affects women following a mastectomy and is referred to as Post Mastectomy Pain Syndrome (PMPS). Regional anesthesia utilizing single dose nerve blocks is frequently utilized in the preoperative period for many surgical procedures and decreases postoperative pain. Regional anesthesia also frequently results in decreased narcotic use in the post-operative period. The use of regional fascial plane blocks or Pectoralis (PECs) blocks has increased in the setting of mastectomy. The regional block utilizes ultrasound guidance to inject local anesthesia into the fascial planes of muscles thereby infiltrate the surrounding nerves. One example is the pectoral I block which deposits local anesthetic between the pectoralis major and minor muscles and pectoral II above the serratus anterior muscle with an intended blockade for intercostals III, IV, V, VI and long thoracic nerves. These techniques have shown a decrease in postoperative pain and postoperative narcotic consumption. The investigators seek to evaluate if preoperative regional nerve blocks decrease post mastectomy chronic pain, improving the quality of life of breast cancer survivors. Therefore, the aim of this study is to determine whether regional nerve blocks affect chronic post-mastectomy pain and whether the regional block is associated with perioperative pain and postoperative narcotic consumption.

ELIGIBILITY:
Inclusion Criteria:

1. Women at least 19 years old who are able to provide written and informed consent
2. Women undergoing unilateral or bilateral, simple, skin-sparing, or nipple sparing mastectomy for breast cancer (Stage 0-III) or breast cancer prevention
3. Patients with ASA class of I-III will be included

Exclusion Criteria:

1. Stage IV breast cancer, morbid obesity with BMI >45kg/m2
2. Renal insufficiency (Creatinine >1.5 mg/dL)
3. Current chronic analgesic use (daily use for > or equal to 4 weeks)
4. History of opioid abuse or dependence
5. Presence of chronic pain with a self-reported average pain score of 4 or greater on a pain scale of 0-10 prior to any surgical intervention
6. Incarceration
7. Pregnancy
8. Immediate autologous tissue reconstruction.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing unilateral or bilateral, simple, skin-sparing, or nipple sparing mastectomy for breast cancer (Stage 0-III) or breast cancer prevention, at least 19 years old, who are able to provide written and informed consent.
Enrollment: 21 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain: Brief Pain Inventory- Short Form (BPI-SF) | Baseline (day of surgery) to 8 hours
  Severity of postoperative pain will be evaluated by the Brief Pain Inventory- Short Form (BPI-SF). This form asks a series of 9 questions with ratings of pain from 0 (no pain) to 10 (pain as severe as you can imagine) and includes questions evaluating general activities of daily living. The study team will evaluate patient reported levels of pain at 8 hours. This series of questions will be administered in person during the inpatient stay and by telephone or in the clinic setting after discharge.
Postoperative Pain | Baseline (day of surgery) to 16 hours (+/- 4 hours)
  Severity of postoperative pain will be evaluated by the Brief Pain Inventory- Short Form (BPI-SF). This form asks a series of 9 questions with ratings of pain from 0 (no pain) to 10 (pain as severe as you can imagine) and includes questions evaluating general activities of daily living. The study team will evaluate patient reported levels of pain at 16 hours (+/- 4 hours). This series of questions will be administered in person during the inpatient stay and by telephone or in the clinic setting after discharge.
Postoperative Pain: Brief Pain Inventory- Short Form (BPI-SF) | Baseline (day of surgery) to 2 days
  Severity of postoperative pain will be evaluated by the Brief Pain Inventory- Short Form (BPI-SF). This form asks a series of 9 questions with ratings of pain from 0 (no pain) to 10 (pain as severe as you can imagine) and includes questions evaluating general activities of daily living. The study team will evaluate patient reported levels of pain at 2 days. This series of questions will be administered in person during the inpatient stay and by telephone or in the clinic setting after discharge.
Postoperative Pain: Brief Pain Inventory- Short Form (BPI-SF) | Baseline (day of surgery) to 14 days (+/- 3 days)
  Severity of postoperative pain will be evaluated by the Brief Pain Inventory- Short Form (BPI-SF). This form asks a series of 9 questions with ratings of pain from 0 (no pain) to 10 (pain as severe as you can imagine) and includes questions evaluating general activities of daily living. The study team will evaluate patient reported levels of pain at 14 days (+/- 3 days). This series of questions will be administered in person during the inpatient stay and by telephone or in the clinic setting after discharge.
Postoperative Pain: Brief Pain Inventory- Short Form (BPI-SF) | Baseline (day of surgery) to 6 months
  Chronic pain will be evaluated by the Brief Pain Inventory- Short Form (BPI-SF). This form asks a series of 9 questions with ratings of pain from 0 (no pain) to 10 (pain as severe as you can imagine) and includes questions evaluating general activities of daily living. The study team will evaluate patient reported levels of pain at 6 months. This series of questions will be in the clinic setting after discharge.
Postoperative Pain: Brief Pain Inventory- Short Form (BPI-SF) | Baseline (day of surgery) to 12 months
  Chronic pain will be evaluated by the Brief Pain Inventory- Short Form (BPI-SF). This form asks a series of 9 questions with ratings of pain from 0 (no pain) to 10 (pain as severe as you can imagine) and includes questions evaluating general activities of daily living. The study team will evaluate patient reported levels of pain at 12 months. This series of questions will be in the clinic setting after discharge.

SECONDARY OUTCOMES:
Postoperative narcotic consumption | Baseline (day of surgery) to discharge (approximately 2 to 30 days post surgery)
  Post-operative narcotic consumption will be measured as the total number of oral morphine-equivalent units administered during hospitalization and subsequent narcotic use will be patient-reported narcotic consumption which will also be converted into oral morphine.
Postoperative nausea | Baseline (day of surgery) to 48 hours after surgery
  Patient self-reported nausea within 48 hours after surgery.
Postoperative length of stay | Baseline (day of surgery) to discharge (approximately 2 to 30 days post surgery)
  Total length of patients hospital stay after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Rachael B Lancaster, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Hospitals and Affiliated Clinics, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No